CLINICAL TRIAL: NCT05089123
Title: Prospective, Multicenter, Double-blind, Randomized, Comparative Immunogenicity and Safety Trial of Flu-M [Inactivated Split Influenza Vaccine], Solution for Intramuscular Injection, 0.5 ml (FSUE SPbSRIVS FMBA), vs. Ultrix®, Solution for Intramuscular Injection, 0.5 ml (FORT LLC) in Volunteers Aged Over 60 Years
Brief Title: The Objectives of This Study Are Study the Immunogenicity and Safety of the Flu-M [Inactivated Split Influenza Vaccine], vs. the Ultrix® Inactivated Split Influenza Vaccine, in Volunteers Who Are Over 60 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FM-2019-02
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-10

CONDITIONS: Influenza
Keywords: influenza; flu; vaccine; Flu-M
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flu-M (Experimental): 160 volunteers were vaccinated with the Flu-M inactivated split influenza vaccine with a preservative
  Interventions: Biological: Flu-M [Inactivated split influenza vaccine]
- Ultrix (Active Comparator): 160 volunteers were vaccinated with the Ultrix (Inactivated split influenza vaccine)
  Interventions: Biological: Inactivated Split Influenza Vaccine

INTERVENTIONS:
Biological: Flu-M [Inactivated split influenza vaccine] — solution for intramuscular injection, 0.5 ml
  Arms: Flu-M
Biological: Inactivated Split Influenza Vaccine — solution for intramuscular injection, 0.5 ml
  Arms: Ultrix

SUMMARY:
This trial by its design was a prospective, multicenter, double blind, randomized comparative clinical trial of the IIIb-IV phase which was carried out in parallel groups of volunteers over the age of 60

DETAILED DESCRIPTION:
The volunteers will include in the trial will divide into two groups:

Group 1: volunteers who will receive one dose of Flu-M, solution for intramuscular injection, 0.5 mL, intramuscularly.

Group 2: volunteers who will receive one dose of Ultrix®, solution for intramuscular administration, 0.5 mL, intramuscularly.

The trial include the following periods and visits:

1. Screening period (up to 7 days):

   • Visit 0 (day -7...-1).
2. Vaccination period (up to 1 day):

   • Visit 1 (day 1, randomization, blood collection for serological examination, vaccination).
3. Follow-up period (up to 28(+2) days):

   * Visit 2 (day 3, organization of trials to assess safety);
   * Visit 3 (day 7(+1), organization of trials to assess safety);
   * Visit 4 (day 21(+2), organization of trials to assess safety, blood collection for serological study);
   * Visit 5 (day 28(+2), organization of trials to assess safety, trial completion);

ELIGIBILITY:
Inclusion Criteria:

* Presence of signed informed consent to participate in the trial.
* Volunteers (both male and female) over the age of 60 who could meet the Protocol requirements.
* Negative pregnancy test obtained from female volunteers with preserved childbearing potential.
* Consent to use adequate contraception methods (contraception methods with degree of reliability of more than 90%: a nonhormonal intrauterine device; a spermicide condom; a spermicide cervical cap; spermicide diaphragms) or total sexual abstinence during the clinical trial (until Visit 5 (day 28(+2)).

Exclusion Criteria:

* Allergic reactions to chicken protein or any previous influenza vaccination.
* Anamnestic data on the episodes of severe allergic reactions and/or diseases (anaphylaxis, Quincke's edema, polymorphic exudative erythema, serum disease etc.)
* Acute reaction (temperature above 38.5оС, edema and hyperemia over 5 cm in diameter at the injection site) or complications caused by previous administration of the drug.
* Previous vaccination 6 months before the start of the trial.
* History of leucosis, blood cancer, malignant oncological diseases.
* Guillain-Barré syndrome (acute polyneuropathy) in the medical history.
* Positive screening for HIV infection, B and C hepatitis, syphilis.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition;
* Administration of immunoglobulin or blood products within the last three months before the study.
* Long-term use (more than 14 days) of immunosuppressants (including systemic corticosteroids, cytotoxic, radioactive preparations) or other immunomodulatory drugs for six months before the trial.
* Chronic diseases at the decompensation stage or in debilitating form, which can make it dangerous for the volunteer to take part in the trial.
* Progressive neurological disorders, dementia.
* Blood disorders which serve as a contradiction for intramuscular injection.
* History of alcohol or drug addiction.
* Pregnancy, breastfeeding in women with preserved reproductive performance.
* Current participation in another clinical trial or within the previous 3 months before the screening.
* Mental, physical and other problems which do not allow for appropriate assessment of own behavior and following the requirements set out in the trial protocol.
* Any other conditions which in the reasonable opinion of the clinical investigator complicate the participation of the volunteer in the trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Immunogenicity assessment | 21 days
  Seroconversion rate defined as the percentage of subjects who have a pre-vaccination titer of influenza haemagglutinin antibody titer (HA titer) < 1:10 and a post-vaccination HA titer >1:40 or a pre-vaccination HA titer > 1:10 and at least a fourfold increase in post-vaccination HA titer vs. the baseline for each strain (A/H1N1, A/H3N2 and B)

SECONDARY OUTCOMES:
The percentage of subjects with protective titer of antibodies ≥ 1:40 on the 21(+2) day after the vaccination for each strain (A/H1N1, A/H3N2 and B). | 21 days
Increasing of geometric mean titer on the 21(+2) day against the value observed before the use of vaccine for each strain (A/H1N1, A/H3N2 and B) | 21 days
The percentage of volunteers with a pre-vaccination HA titer <1:10 and a post-vaccination HA titer >1:40 or a pre-vaccination HA titer > 1:10 and at least a fourfold increase in a post-vaccination HA titer vs. the baseline should be > 30% | 21 days
Increasing of geometric mean titer in > 2.0 times | 21 days
The percentage with protective antibody titer ≥ 1:40 | 21 days

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - LLC "Meditsinskie Tehnologii", Saint Petersburg
  - LLC "Strategicheskie Meditsinskie Sistemi", Saint Petersburg